CLINICAL TRIAL: NCT00172341
Title: Efficacy and Safety of Sublingual Immunotherapy With House Dust Mite Extract in Asthmatic Children: A Double-Blind, Randomized, and Placebo-Controlled Study
Brief Title: Sublingual Immunotherapy With House Dust Mite Extract in Asthmatic Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 930309
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-03 (Estimated); Status verified 2004-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: Staloral TM

SUMMARY:
Asthma, the airway inflammatory disorder, is an important chronic disease in children. About 10~15% children are bothered with this. Allergens, such as house-dust mites (HDM), animal dander (i.e. cats and dogs), and seasonal pollens, are often implicated as causative and triggering factors of respiratory attacks in children with asthma. Among them, mites are the most common indoor allergen associated with asthma worldwide.

It appears that SLIT is somewhat effective and safe. However, on the current evidence, further studies are needed to define the indications, the duration of treatment and therapeutic optimal dose of standardized allergen extracts in relation to efficacy and side effects before it is recommended for routine clinical use. The objective of the present study was to investigate the effects and safety of StaloralTM, the standardized extracts of D. pt. and D. f., in asthmatic children allergic to HDM.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 5 to 15 years; either sex· Patients with asthma at least one year of clinical history and with sensitization to domestic mites, the skin (prick test) tested positive to D. pt. and D. f. showing wheal ³ 5mm, and with specific D. pt. IgE rate ³ Class 4+ when tested by CAP System· Patients with at least 1-year history of mild to moderate of severity of asthma [Steps 2 and 3 GINA (global initiative for asthma)]A) Mild persistent asthma (Step 2 GINA), characterized by - Symptoms: > 2 times per week but < 1 time per day- Exacerbations: Affect activity and sleep - Night-time asthma symptom: > 2 times per month- PEF (peak expiratory flow) or FEV1 (forced expiratory volume in the first second)- ³ 80% predicted- variability 20-30%B) Moderate persistent asthma (Step 3 GINA), characterized by- Symptoms: Daily- Exacerbations: Affect activity and sleep- Night-time asthma symptom: > 1 time per week- PEF or FEV1 - 60 < but < 80% predicted- variability > 30%Reversibility of PEFR (peak expiratory flow rate) ³ 15% after inhaled b2-agonists· Patients or parents who have given informed consent· Patients with a FEV1 greater than 70% of predicted· Patients without hypersensitivity to any other airborne allergens in the standardized prick test panel except house dust mites

Exclusion Criteria:

* Perennial allergenic asthma and co-sensitization to Cockroach, Alternaria or Cladosporium, dog and/or cat dander and seasonal asthma due to pollens. The co-sensitization involved are established by: - Pertinent clinical history- Positive skin prick test (wheal ³5mm)- Specific IgE rate ³2+ (tested by CAP)· Patients have been treated by subcutaneous immunotherapy with D. pt. and D. f. mites in the past 2 years· Patients with contraindication to specific-allergen immunotherapy, such as immunodepression, autoimmune diseases, progressive nephropathy and malignancy of any system· Patients with peptic ulcers, reflux-esophagitis and other conditions such as ulcer/erosion proved by upper gastroenteric endoscopy or the history of upper gastroenteric tract bleeding· Patients with anatomical abnormality of upper respiratory tracts· Patients with atopic dermatitis · Patients participating in other clinical trials within the past 3 months prior to the study· Patients with any form administration of immunotherapy in previous years or ongoing· Patients with a history of cardiovascular, psychotic or other medical or immunologic diseases· Patients with other active pulmonary diseases such as tuberculosis, pneumonia or pulmonary edema· Patients who were treated with oral or parenteral corticosteroids (more than 15 consecutive days), depot steroids, inhaled corticosteroids in a dosage greater than 1000 mg/day (beclomethasone dipropionate), inhaled b2-agonists more than four times daily and/or oral b2-agonists or methylxanthines· Female patients who are pregnant, nursing or childbearing potential are not included.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100

PRIMARY OUTCOMES:
Change of asthmatic scores from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Li-Chieh Wang, MD, Principal Investigator — National Taiwan University Hospital